CLINICAL TRIAL: NCT01826305
Title: Independent Exercise Compared With Formal Rehabilitation Following Primary Total Knee Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-09642
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Recovery Following Primary Total Knee Arthroplasty
MeSH Terms: interventions — Physical Therapy Modalities

ARMS (2):
- Formal Rehabilitation Therapy (Active Comparator): Patients randomized to the formal rehabilitation therapy cohort will receive a prescription for therapy for twelve weeks following their primary knee replacement.
  Interventions: Procedure: Formal Rehabilitation Therapy
- Independent Exercise Cohort (Experimental): Patients randomized to the independent exercise cohort will receive online access to a twelve-week protocol of exercises to perform at home to strengthen and improve function of the replaced knee.
  Interventions: Procedure: Independent Exercise Cohort

INTERVENTIONS:
Procedure: Formal Rehabilitation Therapy — Patients that will be randomized to the formal rehabilitation therapy cohort will be prescribed formal therapy for twelve weeks with supervised exercises to regain knee strength and range of motion. Therapists will not be involved in the study design and therapists will not be informed that patients are participating in this study. The content, frequency, and duration of the rehabilitation program will be at the discretion of the treating therapist, consistent with usual practice.
  Other Names: Physical Therapy
  Arms: Formal Rehabilitation Therapy
Procedure: Independent Exercise Cohort — The patients who will be in the independent exercises cohort will be registered on www.careforpatients.com, an online rehabilitation resource that provides computer aided rehabilitative exercises. Patients will follow a prepared 12-week protocol of exercises to perform post-operatively to gradually regain their knee strength, flexion, extension, abduction, and adduction.
  Arms: Independent Exercise Cohort

SUMMARY:
In this study we plan to compare the efficacy of independent exercises performed by the patients at home to formal rehabilitation therapy following primary total knee replacement. Patients will be randomized to these two cohorts at enrollment into the study and followed prospectively. Patients randomized to the formal rehabilitation cohort will receive a prescription for therapy for twelve weeks. Patients randomized to the independent exercise cohort will receive online access to a twelve-week protocol of exercises to perform at home to strengthen and improve function of the replaced joint.

At enrollment, a baseline evaluation will be conducted to capture demographics, height, weight, primary diagnosis, medical comorbidities, and social supports as well as completion of the selected outcome measure, American Knee Society (AKS) Score, Knee and Osteoarthritis Outcome Score (KOOS). Secondary outcomes will include the measurement of health status with use of the Short Form-12v2 (SF-12v2) and activity level with the University of California, Los Angeles (UCLA) Activity Score. At the twelve-week, six-month and twelve-month follow-up visits, the study subjects will complete the KOOS, SF-12v2, and UCLA Activity Score questionnaires. Statistical analysis will be performed to compare the outcomes between the two cohorts.

Hypothesis:

There will be no difference in outcomes between formal rehabilitation and independent exercises at twelve months after primary total knee replacement surgery using the American Knee Society (AKS) Knee Score.

DETAILED DESCRIPTION:
We will randomize patients who are scheduled to have primary total knee arthroplasty to receive either a prescription for formal physical therapy (PT) or instructions for independent exercises. Inclusion criteria will be: scheduled for primary total knee arthroplasty, an age of eighteen years or older, speak English, and have a computer with access to the Internet. Exclusion criteria will be: any knee arthroplasty other than total knee, patients not planning to return for follow up care, patients relying on others for basic functioning, do not speak English, and do not have a computer with access to the Internet. Enrollment will occur at the initial clinic visit in the surgeon's office.

Informed consent will be received from patients who will participate in the study at the initial clinic visit and these patients will be randomized equally to either the PT/OT or independent exercise cohort using the REDCap website randomization feature. REDCap is a secure, web-based application for building and managing online surveys and databases that will be utilized for this study for data management. Patients that will be randomized to PT cohort will be prescribed formal therapy for twelve weeks with supervised exercises to regain knee strength and range of motion. Therapists will not be involved in the study design and therapists will not be informed that patients are participating in this study. The content, frequency, and duration of the rehabilitation program will be at the discretion of the treating therapist, consistent with usual practice.

The patients who will be in the independent exercises cohort will be registered on www.careforpatients.com, an online rehabilitation resource that provides computer aided rehabilitative exercises. Patients will follow a prepared 12-week protocol of exercises to perform postoperatively to gradually regain their knee strength and range of motion.

Post-operative weeks 0 - 1, the patients will perform three sets of ten repetitions everyday of: supine ankle pumps, supine heel slides, seated quad sets, supine glut sets, and supine hip abduction/adduction. The patient will also perform three sets of patella mobilization for one minute each and three sets of one repetition of supine knee extension.

Post-operative weeks 1 - 2, the patients will perform three sets of ten repetitions everyday of: supine heel slides, prone knee flexion, supine knee extension, supine SLR flexion, sidelying SLR abduction, prone SLR extension, sidelying SLR adduction. The patient will also perform three sets of patella mobilization for one minute each and three sets of one repetition of supine knee extension with weight.

Post-operative weeks 2 - 4, the patients will perform three sets of ten repetitions everyday of: standing knee extension, standing knee flexion, standing SLR flexion, standing SLR abduction, standing SLR extension, standing SLR adduction. The patient will also perform three sets of patella mobilization for one minute each, three sets of sitting hamstring stretch for thirty seconds each, prone quad stretch for thirty seconds each, and three sets of single leg stance for thirty seconds each.

Post-operative weeks 4 - 8, the patients will perform three sets of ten repetitions everyday of: bilateral mini squats, standing SLR flexion, standing SLR abduction, standing SLR extension, standing SLR adduction. The patient will also perform three sets of sitting hamstring stretch for thirty seconds each and prone quad stretch for thirty seconds each.

Post-operative weeks 8 - 12, the patients will perform three sets of ten repetitions everyday of: bilateral wall squats, forward step-ups, and side step-ups. The patient will also perform three sets of sitting hamstring stretch for thirty seconds each and prone quad stretch for thirty seconds each. Patients will be advised to perform these exercises as often as possible, but at least once a day.

All patients will have regularly scheduled follow-up visits per usual practice at six-weeks post-operatively, six-months post-operatively, and 12-months post-operatively where a physical exam will be performed to check the range of motion of the knee, gait, and lower leg muscle strength.

The primary outcome of the trial will be to evaluate the efficacy of formal therapy compared with independent exercises at twelve months after surgery with use of the American Knee Society (AKS) Knee Score. Secondary outcomes will include the Knee and Osteoarthritis Outcome Score (KOOS) the measurement of health status with use of the Short Form-12v2 (SF-12v2) and activity level with the University of California, Los Angeles (UCLA) Activity Score.

At enrollment, a baseline evaluation will be conducted to capture demographics, height, weight, primary diagnosis, medical comorbidities, and social supports as well as completion of the selected outcome measures, AKS, KOOS, SF-12v2, and UCLA Activity Score. At the twelve-week, six-month and twelve-month follow-up visits, the study subjects will complete the AKS, KOOS, SF-12v2, and UCLA Activity Score questionnaires during their clinic visit or will be contacted by telephone or mail to complete the questionnaires if they do not have appointments for twelve-week, six-month or twelve-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for primary total knee arthroplasty
* an age of eighteen years or older
* English speaking
* have a computer with access to the Internet

Exclusion Criteria:

* any knee arthroplasty other than total knee
* patients not planning to return for follow up care
* patients relying on others for basic functioning
* do not speak English
* do not have a computer with access to the Internet
* prior physical therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-07; Primary Completion 2015-10-23 (Actual); Study Completion 2015-10-23 (Actual)

PRIMARY OUTCOMES:
Knee Function | up to 12 months post-operatively
  The American Knee Society Score (AKS) consists of two parts. The first is the Knee Score, which considers pain, stability and range of motion as the main parameters, with deductions for flexion contractures, extension lag and malalignment. The second part, the Function Score, utilizes walking distance and stair climbing as the main parameters with deductions for the use of a walking aid.

SECONDARY OUTCOMES:
General physical and mental health | up to 12 months post-operatively
  The Short Form 12v2 (SF-12v2) is an abbreviated version of the Short Form-36 (SF-36) that includes the physical and emotional limitations that are placed on work and social activities. The SF-12v2 measures how individuals value their current health state. It has been shown to be reliable (Pearson r > 0.70), valid (highly correlated with SF-36), and responsive for the measurements of health status in many patient populations.
Activity Level | up to 12 months post-operatively
  The UCLA Activity Score assesses an individual's level of activity. The evaluation has ten descriptive activity levels ranging from wholly inactive and dependent on others (level 1), to moderate activities such as unlimited housework and shopping (level 6), to regular participation in impact sports such as jogging or tennis (level 10). The individual is asked to pick the statement that best describes their activity level.
Knee and Osteoarthritis Outcome Score (KOOS) | up to 12 months post-operatively
  The KOOS is a self-administered 40-item questionnaire used to assess patient-relevant outcomes in five separate subscales related to the knee (pain, symptoms, activity of daily living, sport and recreation function and knee related quality of life). The KOOS contains all Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) questions in unchanged form, so a WOMAC score can be calculated from the KOOS. The WOMAC is used to assess pain, function, and stiffness of the knee.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J. Bozic, MD, MBA, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Mahomed NN, Davis AM, Hawker G, Badley E, Davey JR, Syed KA, Coyte PC, Gandhi R, Wright JG. Inpatient compared with home-based rehabilitation following primary unilateral total hip or knee replacement: a randomized controlled trial. J Bone Joint Surg Am. 2008 Aug;90(8):1673-80. doi: 10.2106/JBJS.G.01108. PMID 18676897
- [Background] Khan F, Ng L, Gonzalez S, Hale T, Turner-Stokes L. Multidisciplinary rehabilitation programmes following joint replacement at the hip and knee in chronic arthropathy. Cochrane Database Syst Rev. 2008 Apr 16;2008(2):CD004957. doi: 10.1002/14651858.CD004957.pub3. PMID 18425906
- [Background] Shepperd S, Iliffe S. Hospital at home versus in-patient hospital care. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD000356. doi: 10.1002/14651858.CD000356.pub2. PMID 16034853
- [Background] Mahomed NN, Koo Seen Lin MJ, Levesque J, Lan S, Bogoch ER. Determinants and outcomes of inpatient versus home based rehabilitation following elective hip and knee replacement. J Rheumatol. 2000 Jul;27(7):1753-8. PMID 10914863
- [Background] Shepperd S, Harwood D, Jenkinson C, Gray A, Vessey M, Morgan P. Randomised controlled trial comparing hospital at home care with inpatient hospital care. I: three month follow up of health outcomes. BMJ. 1998 Jun 13;316(7147):1786-91. doi: 10.1136/bmj.316.7147.1786. PMID 9624068
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Dorr LD, Maheshwari AV, Long WT, Wan Z, Sirianni LE. Early pain relief and function after posterior minimally invasive and conventional total hip arthroplasty. A prospective, randomized, blinded study. J Bone Joint Surg Am. 2007 Jun;89(6):1153-60. doi: 10.2106/JBJS.F.00940. PMID 17545416
- [Background] Munin MC, Rudy TE, Glynn NW, Crossett LS, Rubash HE. Early inpatient rehabilitation after elective hip and knee arthroplasty. JAMA. 1998 Mar 18;279(11):847-52. doi: 10.1001/jama.279.11.847. PMID 9515999
- [Background] Nilsdotter AK, Lohmander LS, Klassbo M, Roos EM. Hip disability and osteoarthritis outcome score (HOOS)--validity and responsiveness in total hip replacement. BMC Musculoskelet Disord. 2003 May 30;4:10. doi: 10.1186/1471-2474-4-10. Epub 2003 May 30. PMID 12777182
- [Background] Roos EM, Toksvig-Larsen S. Knee injury and Osteoarthritis Outcome Score (KOOS) - validation and comparison to the WOMAC in total knee replacement. Health Qual Life Outcomes. 2003 May 25;1:17. doi: 10.1186/1477-7525-1-17. PMID 12801417
- [Background] Nilsdotter AK, Toksvig-Larsen S, Roos EM. A 5 year prospective study of patient-relevant outcomes after total knee replacement. Osteoarthritis Cartilage. 2009 May;17(5):601-6. doi: 10.1016/j.joca.2008.11.007. Epub 2008 Nov 21. PMID 19091604
- [Background] Hurst NP, Ruta DA, Kind P. Comparison of the MOS short form-12 (SF12) health status questionnaire with the SF36 in patients with rheumatoid arthritis. Br J Rheumatol. 1998 Aug;37(8):862-9. doi: 10.1093/rheumatology/37.8.862. PMID 9734677
- [Background] Terwee CB, Bouwmeester W, van Elsland SL, de Vet HC, Dekker J. Instruments to assess physical activity in patients with osteoarthritis of the hip or knee: a systematic review of measurement properties. Osteoarthritis Cartilage. 2011 Jun;19(6):620-33. doi: 10.1016/j.joca.2011.01.002. Epub 2011 Jan 18. PMID 21251989
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Collins NJ, Misra D, Felson DT, Crossley KM, Roos EM. Measures of knee function: International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form, Knee Injury and Osteoarthritis Outcome Score (KOOS), Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS), Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL), Lysholm Knee Scoring Scale, Oxford Knee Score (OKS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Activity Rating Scale (ARS), and Tegner Activity Score (TAS). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S208-28. doi: 10.1002/acr.20632. No abstract available. PMID 22588746